CLINICAL TRIAL: NCT06836076
Title: Assessment of Depression, Anxiety and ADHD Among Children and Adolescents with Congenital Heart Disease.
Acronym: Psychiatricy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samia Ashraf Abbdelgawad, resident doctor, Assiut University
Other Study IDs: Psychiatric disorders children
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Assessment of Depression, Anxiety and ADHD Among Children and Adolescents with Congenital Heart Disease
Keywords: congenital heart disease; Assessment of depression, anxiety and ADHD
MeSH Terms: conditions — Anxiety Disorders; Heart Defects, Congenital; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Congenital heart disease (CHD) is the most common birth defect, affecting ∼1% of all live births.The spectrum of CHD is wide, ranging from simple (not requiring immediate or possibly any surgical intervention) to severe or complex (typically defined as CHD requiring surgical intervention within the first month to year of life).

DETAILED DESCRIPTION:
Although overall mortality has improved, most notably in those with complex CHD, many surgical and medical procedures are palliative, and these patients often require multiple interventions throughout their lifetime. Increased CHD survival is now resulting in a continually growing population of adolescents and adults with CHD; this has drawn more attention to the noncardiac comorbidities, including overall mental health, of patients with CHD.There are multiple psychological theories that can potentially explain some of the mental health disorders seen in patients with CHD, such as stressful life events and sociocultural impacts (eg, parenting style).Cognitive models, including learned helplessness and negative information processing, may also contribute to the mental health of children with CHD, who often spend significant amounts of time in the hospital and undergo cardiac procedures and surgeries. The presence of underlying genetic syndromes, parental mental health disorders, cardiopulmonary bypass, prematurity, and prolonged hospitalizations are factors that increase the risk of neurodevelopmental disabilities (NDDs) and likely contribute to anxiety, depression, and attention-deficit/hyperactivity disorder (ADHD) in adolescents and adults with complex CHD.

ELIGIBILITY:
Inclusion Criteria:

* childern age from 6 to less than 18
* childern with simple and complex CHD
* in patient and out patient childern
* preoperative and postoperative patient

Exclusion Criteria:

* patient indicated for icu
* patient with critical arrythmias
* caregiver refuse to participate in the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: depression, anxiety and ADHD among children and adolescents with congenital heart disease.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
• The Child Behaviour Checklist (CBCL/6-18) (arabic version) | 1 years
  is a 113-item parent report measure designed to assess behavioural and emotional problems in children and young people aged 6-18 years. This most recent version of the original measure includes items and subscales aimed at assessing symptoms of anxiety, depression, somatic complaints (that is, physiological symptoms frequently associated with internalising behaviours like anxiety and depression), social problems, thought problems, attention problems, rule-breaking behaviour and aggressive behaviour.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bernaras E, Jaureguizar J, Garaigordobil M. Child and Adolescent Depression: A Review of Theories, Evaluation Instruments, Prevention Programs, and Treatments. Front Psychol. 2019 Mar 20;10:543. doi: 10.3389/fpsyg.2019.00543. eCollection 2019. PMID 30949092